CLINICAL TRIAL: NCT00689871
Title: Safety and Effectiveness of Natrelle(TM) Cohesive Round Silicone-Filled Breast Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 020056
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-01

CONDITIONS: Breast Augmentation; Breast Reconstruction; Revision of Augmentation or Reconstruction

ARMS (4):
- 1 (Experimental): Primary augmentation
  Interventions: Device: Natrelle(TM) Silicone-Filled Breast Implants
- 2 (Experimental): Primary reconstruction
  Interventions: Device: Natrelle(TM) Silicone-Filled Breast Implants
- 3 (Experimental): Revision-augmentation
  Interventions: Device: Natrelle(TM) Silicone-Filled Breast Implants
- 4 (Experimental): Revision-reconstruction
  Interventions: Device: Natrelle(TM) Silicone-Filled Breast Implants

INTERVENTIONS:
Device: Natrelle(TM) Silicone-Filled Breast Implants — Breast implant surgery

SUMMARY:
Safety and effectiveness of Natrelle™ Cohesive Round Silicone-Filled Breast Implants in women undergoing primary augmentation, primary reconstruction, or revision of existing breast implants.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years or older
* Seeking primary breast augmentation (i.e., no previous breast implant surgery) indicated for the following: patient dissatisfaction with size or shape of breast (e.g., mammary hypoplasia, asymmetry, ptosis, or aplasia
* Seeking primary breast reconstruction
* Seeking breast revision-augmentation
* Seeking breast revision-reconstruction
* Adequate tissue available to cover implants
* Patients at MRI designated sites must be willing to undergo MRI at their 1,3, 5, 7 and 9-year follow-up visits (serial MRI). The patient must be eligible for MRI (for example, no implanted metal or metal devices and no history of severe claustrophobia that may make her ineligible for MRI).

Exclusion Criteria:

* Advanced fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy
* Existing carcinoma of the breast, without mastectomy
* Abscess or infection in the body at the time of enrollment
* Pregnant or nursing
* Have any disease, including uncontrolled diabetes (e.g., HbAIc > 8%), that is clinically known to impact wound healing ability
* Show tissue characteristics that are clinically incompatible with mammaplasty, such as tissue damage resulting from radiation, inadequate tissue, compromised vascularity or ulceration
* Have, or under treatment for, any condition that may constitute an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems)
* Show psychological characteristics that may be incompatible with the surgical procedure and the prosthesis, such as inappropriate attitude or motivation (e.g., body dysmorphic disorder)
* Are not willing to undergo further surgery for revision, if medically required

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 1999-01; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Spear SL, Murphy DK, Slicton A, Walker PS; Inamed Silicone Breast Implant U.S. Study Group. Inamed silicone breast implant core study results at 6 years. Plast Reconstr Surg. 2007 Dec;120(7 Suppl 1):8S-16S. doi: 10.1097/01.prs.0000286580.93214.df. PMID 18090808
- [Result] Gladfelter J, Murphy D. Breast augmentation motivations and satisfaction: a prospective study of more than 3,000 silicone implantations. Plast Surg Nurs. 2008 Oct-Dec;28(4):170-4; quiz 175-6. doi: 10.1097/PSN.0b013e31818ea7e0. PMID 19092580
- [Result] Murphy DK, Beckstrand M, Sarwer DB. A prospective, multi-center study of psychosocial outcomes after augmentation with natrelle silicone-filled breast implants. Ann Plast Surg. 2009 Feb;62(2):118-21. doi: 10.1097/SAP.0b013e31817f01f8. PMID 19158517
- [Result] Largent JA, Reisman NR, Kaplan HM, Oefelein MG, Jewell ML. Clinical trial outcomes of high- and extra high-profile breast implants. Aesthet Surg J. 2013 May;33(4):529-39. doi: 10.1177/1090820X13484035. Epub 2013 Apr 4. PMID 23559355
- [Result] Namnoum JD, Largent J, Kaplan HM, Oefelein MG, Brown MH. Primary breast augmentation clinical trial outcomes stratified by surgical incision, anatomical placement and implant device type. J Plast Reconstr Aesthet Surg. 2013 Sep;66(9):1165-72. doi: 10.1016/j.bjps.2013.04.046. Epub 2013 May 9. PMID 23664574
- [Derived] Spear SL, Murphy DK; Allergan Silicone Breast Implant U.S. Core Clinical Study Group. Natrelle round silicone breast implants: Core Study results at 10 years. Plast Reconstr Surg. 2014 Jun;133(6):1354-1361. doi: 10.1097/PRS.0000000000000021. PMID 24867717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: January 6, 1999-June 30, 2000 at multiple US sites
Groups:
- Primary Augmentation: All women implanted for an indication of primary breast augmentation
- Primary Reconstruction: All women implanted for an indication of primary breast reconstruction
- Revision-augmentation: All women implanted for revision of a breast augmentation
- Revision-reconstruction: All women implanted for revision of a breast reconstruction
Period: Overall Study
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision-augmentation | Revision-reconstruction
Started | 455 (908 Implants) | 98 (127 Implants) | 147 (288 Implants) | 15 (25 Implants)
Completed | 280 (35 Patients discontinued) | 46 (35 Patients discontinued) | 74 (28 Patients discontinued) | 8 (4 Patients discontinued)
Not Completed | 175 | 52 | 73 | 7
Not completed — Lost to Follow-up | 123 | 13 | 37 | 1
Not completed — Explanted of All Study Devices | 36 | 25 | 29 | 3
Not completed — Withdrawal by Subject | 13 | 3 | 4 | 1
Not completed — Death | 1 | 10 | 2 | 2
Not completed — Physician Decision | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision-augmentation | Revision-reconstruction | Total
Number analyzed (Participants) | 455 | 98 | 147 | 15 | 715
Age, Customized [Number; unit: participants]
  <=40 years | 319 | 10 | 61 | 0 | 390
  Between 40 and 60 years | 136 | 73 | 84 | 9 | 302
  >=60 years | 0 | 15 | 2 | 6 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455 | 98 | 147 | 15 | 715
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Local Complications
Description: By patient risk of complications occuring in at least 5% of patients in 1 or more cohorts
Time Frame: 10 years
Population: all enrolled patients
Measure: Number (95% Confidence Interval); unit: percentage by patient
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision-augmentation | Revision-reconstruction
Number analyzed (Participants) | 455 | 98 | 147 | 15
percentage by patient
  Capsular Contracture | 18.9 [15.4 to 23.1] | 24.6 [16.2 to 36.2] | 28.7 [21.3 to 37.9] | 6.7 [0.2 to 31.9]
  Breast Pain | 11.5 [8.7 to 15.0] | 6.8 [2.8 to 16.1] | 11.7 [7.1 to 18.8] | 0 [0 to 0]
  Swelling | 9.2 [6.8 to 12.4] | 7.1 [3.5 to 14.4] | 8.2 [4.6 to 14.5] | 0 [0 to 0]
  Implant Malposition | 6.9 [4.8 to 9.7] | 2.3 [0.6 to 8.9] | 6.0 [3.1 to 11.7] | 13.3 [1.7 to 40.5]
  Nipple Complications | 6.3 [4.3 to 9.1] | 3.3 [1.1 to 9.8] | 1.4 [0.3 to 5.4] | 0 [0 to 0]
  Hypertrophic/Other Abnormal Scarring | 4.2 [2.6 to 6.5] | 5.5 [2.3 to 12.7] | 6.6 [3.5 to 12.3] | 0 [0 to 0]
  Asymmetry | 3.3 [2.0 to 5.6] | 23.2 [15.4 to 33.9] | 6.5 [3.2 to 12.8] | 6.7 [0.2 to 31.9]
  Wrinkling | 1.8 [0.8 to 3.7] | 10.2 [5.2 to 19.6] | 5.4 [2.6 to 11.0] | 0 [0 to 0]
  Implant Palpability/Visibility | 1.6 [0.8 to 3.4] | 6.4 [2.3 to 12.7] | 6.0 [3.0 to 11.6] | 6.7 [0.2 to 31.9]
  Seroma/Fluid Accumulation | 1.8 [0.9 to 3.4] | 2.3 [0.3 to 15.4] | 6.0 [3.0 to 11.6] | 6.7 [0.2 to 31.9]
  Bruising | 0.4 [0.1 to 1.8] | 1.0 [0.1 to 7.1] | 3.0 [1.1 to 7.8] | 6.7 [0.2 to 31.9]
  Skin Rash | 0.9 [0.3 to 2.3] | 2.0 [0.5 to 7.9] | 0.7 [0.1 to 4.9] | 6.7 [0.2 to 31.9]

2. Secondary Outcome: Satisfaction With Breast Implants as Determined by Patients and Physicians on a 5-point Scale
Description: Satisfaction score on a 5-point scale, where 1 is definitely dissatisfied and 5 is definitely satisfied
Time Frame: 10 years
Population: All patients who had a breast implant satisfaction rating
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision-augmentation | Revision-reconstruction
Number analyzed (Participants) | 279 | 44 | 74 | 8
units on a scale
  Physician satisfaction | 4.8 (0.7) | 4.7 (0.6) | 4.4 (1.1) | 4.6 (1.1)
  Patient satisfaction | 4.8 (0.7) | 4.6 (0.7) | 4.4 (1.2) | 4.5 (1.4)

ADVERSE EVENTS:
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision-augmentation | Revision-reconstruction
Serious Adverse Events (participants affected / at risk) | 0/455 | 0/98 | 0/147 | 0/15
Other Adverse Events (participants affected / at risk) | 0/455 | 0/98 | 0/147 | 0/15

LIMITATIONS AND CAVEATS:
The Revision-reconstruction arm only had 15 patients enrolled, which makes the data for that arm difficult to interpret.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The timing of separate presentation or publication of the study by the PI is subject to mutual agreement in advance between the Sponsor and PI.